CLINICAL TRIAL: NCT01197690
Title: Association Between Fractional Exhaled Nitric Oxide and Asthma Control
Acronym: FeNO_AS
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Other Study IDs: 602/2552(EC1)
Record Dates: First submitted 2010-07-18; First posted 2010-09-09 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; level of control of asthma; fractional exhaled nitric oxide (FeNO); asthma control test (ACT)
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine mean or median of fractional exhaled nitric oxide (FeNO) in Thai atopic asthmatic patients that divided into subgroups due to level of asthma control according to the global initiative for asthma guideline.

DETAILED DESCRIPTION:
From many previous studies, fractional exhaled nitric oxide (FeNO) has many benefits such as non-invasive, easily to perform, less time consume, has direct association with severity of inflammation of bronchial trees and sputum eosinophils, has benefit for diagnosis and monitoring the treatment in asthmatic patients.

In Thailand, this field of study is less extend, especially in children population. We hypothesized that in uncontrolled or partly controlled group may have high level of fractional exhaled nitric oxide (FeNO) than controlled group.

It is therefore desirable to examine the association between fractional exhaled nitric oxide (FeNO) and level of asthma control among atopic asthmatic Thai children and will be the main objective of this research.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of atopic bronchial asthma
* follow up in clinic of allergy and clinical immunology, Siriraj hospital

Exclusion Criteria:

* smoker or past history of smoking
* has chronic disease eg. HIV infection, pulmonary hypertension, systemic lupus erythematosus, liver cirrhosis, gastroesophageal reflux, COPD, bronchiectasis
* drink ethanol within 48 hours before enrollment
* history of upper or lower respiratory tract infection within 6 weeks before enrollment
* drink caffeine within day before enrollment
* during pregnancy
* history of systemic steroid use within 8 weeks before enrollment

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: atopic asthmatic patients in Department of Pediatrics, Siriraj hospital (tertiary care)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
fractional exhaled nitric oxide level | 10 minutes (average time), on the day of enrollment

SECONDARY OUTCOMES:
scores of asthma control test: ACT | 5 minutes (average time), on the day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Nualanong Visitsunthorn, MD, Principal Investigator — Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Thailand